CLINICAL TRIAL: NCT06981572
Title: Comparison of the Effectiveness of Implementing Modified ERAS Protocols vs. Standard Management in Pediatric Patients Undergoing Major Gastrointestinal Surgery
Brief Title: Comparing the Effectiveness of Modified ERAS Protocols vs. Standard Management in Pediatric Gastrointestinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Andi Ade Wijaya Ramlan, Head of Department of Anesthesiology and Intensive Therapy, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IndonesiaUAnes2809
Record Dates: First submitted 2024-03-28; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Surgery; Anesthesia
Keywords: enhanced recovery after surgery; major intestinal surgery

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- modified ERAS protocol applied (Active Comparator): patients modified ERAS protocol applied
  Interventions: Procedure: Modified Enhanced Recovery After Surgery Protocol
- standart protocol applied (No Intervention): patients with standart protocol applied

INTERVENTIONS:
Procedure: Modified Enhanced Recovery After Surgery Protocol — This study is to determine the comparison of the effectiveness of the ERAS modification protocol with the standard protocol in reducing length of stay and improving postoperative outcomes for pediatric patients at RSCM who underwent major gastrointestinal surgery using the ERAS modification method. This study is a single-blind clinical trial. Research subjects will be randomly divided into two groups, namely the group who underwent surgery with the ERAS modification protocol and the group who underwent surgery without the ERAS modification protocol. Modified ERAS protocol will be applied during perioperative
  Arms: modified ERAS protocol applied

SUMMARY:
Perioperative management of pediatric patients with gastrointestinal diseases involves a fairly length process and which can lead to rapid deterioration even death. Preoperative management includes preoperative fasting for such a long time, usage of drains and tubes and post-operative bed rest for a long time which can cause pain, stress, and slowing down the recovery time for normal bowel function, thus further prolonging the patient's stay in hospital. Enhanced recovery after surgery (ERAS) is a concept that seeks faster recovery times for pediatric patients and shortens the length of hospital stay while still improving postoperative outcomes. The ERAS modification protocol aims to optimize inpatient care and minimize patient discomfort. Studies show that implementing the modified ERAS protocol can reduce the duration of hospitalization and the incidence of postoperative complications as well as speedy recovery. However, currently the standard ERAS protocol is difficult to apply to pediatric patients. This study will determine the comparison of the effectiveness of the ERAS modification protocol with the standard protocol in reducing length of stay and improving postoperative outcomes for pediatric patients at RSCM who underwent major gastrointestinal surgery using the ERAS modification method.

DETAILED DESCRIPTION:
Perioperative management of pediatric patients with gastrointestinal diseases involves a fairly length process and which can lead to rapid deterioration even death. Preoperative management includes preoperative fasting for such a long time, usage of drains and tubes and post-operative bed rest for a long time which can cause pain, stress, and slowing down the recovery time for normal bowel function, thus further prolonging the patient's stay in hospital. Enhanced recovery after surgery (ERAS) is a concept that seeks faster recovery times for pediatric patients and shortens the length of hospital stay while still improving postoperative outcomes. ERAS was first introduced by a Danish surgeon, Henrik Kehlet in the 1990s to reduce perioperative stress and organ dysfunction in surgical patients. ERAS is an evidence-based technique and combines and optimizes various multidisciplinary methods used in conventional surgical management, includes surgery, anesthesia, nursing, and nutrition. ERAS emphasizes perioperative preparation including preoperative counseling, limited time in preoperative fasting, optimal anesthesia, minimally invasive techniques, immediate postoperative oral nutrition and mobilization, and non-routine use of drainage and surgical tubes. The ERAS modification protocol aims to optimize inpatient care and minimize patient discomfort. Studies show that implementing the modified ERAS protocol can reduce the duration of hospitalization and the incidence of postoperative complications as well as speedy recovery. However, currently the standard ERAS protocol is difficult to apply to pediatric patients because several conditions are not possible in pediatric patients, for example, administering anticoagulants, post-operative fasting, etc., thus requiring modifications that are tailored to the characteristics of the patients at Ciptomangunkusumo Hospital. Children experience a more complex surgical stress response than adult patients. Conventional perioperative management in children often results in greater physical stress. Therefore, perioperative management in children needs to be optimized.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 1 month to 2 years
* The patient underwent major gastrointestinal surgery
* ASA 1 and 2 physical status
* The patient will undergo elective lower abdominal surgery with general and regional anesthesia

Exclusion Criteria:

* Patients with cyanotic congenital heart defects
* Patients with metabolic disorders
* Patients with decreased consciousness
* Patients with severe cognitive impairment
* Patients with relaparotomy due to surgical complications

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Length of stay | The timeframe is calculated from when the patient undergoes preoperative assessment until discharge from the hospital, up to 3 months.
  Patients' length of stay in the hospital, measured in days

SECONDARY OUTCOMES:
Blood glucose level (mg/dL) | The time frame includes 1 day before surgery (preoperative), during surgery (intraoperative), and on the 3rd and 5th days after surgery (postoperative)
  Blood glucose levels measured and compared during the preoperative, intraoperative, and postoperative periods
Blood electrolyte levels (Na, K, Cl) | Blood electrolyte levels assessed 1 day before surgery (preoperative) and on the 3rd day after surgery (postoperative)
  Blood electrolyte levels assessed during the preoperative and postoperative periods
Oral Nutrition Initiation Time | The time frame is calculated from the end of the surgery and will be evaluated up to the time of the patient's discharge from the hospital
  The time when the patient begins receiving oral nutrition, starting with clear fluids. Oral nutrition initiation time will be measured in hours
Time to mobilization | The time frame is calculated from the end of surgery and will be evaluated up to the time of the patient's discharge from the hospital
  The time when the patient begins mobilization, which includes turning to the right and left sides, sitting, walking, and eventually resuming preoperative activities without pain or discomfort. The mobilization time is measured in days

CONTACTS AND LOCATIONS:
Overall Officials: Andi Ade Wijaya Ramlan, Study Chair — Anesthesiology and Intensive Therapy Departement
Locations (1):
- Cipto Mangunkusumo Central National Hospital, Jakarta Pusat, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brindle ME, Heiss K, Scott MJ, Herndon CA, Ljungqvist O, Koyle MA; on behalf Pediatric ERAS (Enhanced Recovery After Surgery) Society. Embracing change: the era for pediatric ERAS is here. Pediatr Surg Int. 2019 Jun;35(6):631-634. doi: 10.1007/s00383-019-04476-3. Epub 2019 Apr 25. PMID 31025092
- [Background] Practice Guidelines for Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration: Application to Healthy Patients Undergoing Elective Procedures: An Updated Report by the American Society of Anesthesiologists Task Force on Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration. Anesthesiology. 2017 Mar;126(3):376-393. doi: 10.1097/ALN.0000000000001452. No abstract available. PMID 28045707
- [Background] Smith I, Kranke P, Murat I, Smith A, O'Sullivan G, Soreide E, Spies C, in't Veld B; European Society of Anaesthesiology. Perioperative fasting in adults and children: guidelines from the European Society of Anaesthesiology. Eur J Anaesthesiol. 2011 Aug;28(8):556-69. doi: 10.1097/EJA.0b013e3283495ba1. PMID 21712716
- [Background] Garin C. Enhanced recovery after surgery in pediatric orthopedics (ERAS-PO). Orthop Traumatol Surg Res. 2020 Feb;106(1S):S101-S107. doi: 10.1016/j.otsr.2019.05.012. Epub 2019 Sep 12. PMID 31522902
- [Background] Ceelie I, de Wildt SN, van Dijk M, van den Berg MM, van den Bosch GE, Duivenvoorden HJ, de Leeuw TG, Mathot R, Knibbe CA, Tibboel D. Effect of intravenous paracetamol on postoperative morphine requirements in neonates and infants undergoing major noncardiac surgery: a randomized controlled trial. JAMA. 2013 Jan 9;309(2):149-54. doi: 10.1001/jama.2012.148050. PMID 23299606
- [Background] Carli F. Physiologic considerations of Enhanced Recovery After Surgery (ERAS) programs: implications of the stress response. Can J Anaesth. 2015 Feb;62(2):110-9. doi: 10.1007/s12630-014-0264-0. Epub 2014 Dec 12. PMID 25501695
- [Background] Somri M, Matter I, Parisinos CA, Shaoul R, Mogilner JG, Bader D, Asphandiarov E, Gaitini LA. The effect of combined spinal-epidural anesthesia versus general anesthesia on the recovery time of intestinal function in young infants undergoing intestinal surgery: a randomized, prospective, controlled trial. J Clin Anesth. 2012 Sep;24(6):439-45. doi: 10.1016/j.jclinane.2012.02.004. Epub 2012 Jul 2. PMID 22762977
- [Background] Narvey MR, Marks SD. The screening and management of newborns at risk for low blood glucose. Paediatr Child Health. 2019 Dec;24(8):536-554. doi: 10.1093/pch/pxz134. Epub 2019 Dec 9. PMID 31844395
- [Background] Gao R, Yang H, Li Y, Meng L, Li Y, Sun B, Zhang G, Yue M, Guo F. Enhanced recovery after surgery in pediatric gastrointestinal surgery. J Int Med Res. 2019 Oct;47(10):4815-4826. doi: 10.1177/0300060519865350. Epub 2019 Aug 4. PMID 31379230
- [Background] George JA, Salazar AJG, Irfan A, Prichett L, Nasr IW, Garcia AV, Boss EF, Jelin EB. Effect of implementing an enhanced recovery protocol for pediatric colorectal surgery on complication rate, length of stay, and opioid use in children. J Pediatr Surg. 2022 Jul;57(7):1349-1353. doi: 10.1016/j.jpedsurg.2022.01.004. Epub 2022 Jan 15. PMID 35153077
- [Background] Phillips MR, Adamson WT, McLean SE, Hance L, Lupa MC, Pittenger SL, Dave P, McNaull PP. Implementation of a pediatric enhanced recovery pathway decreases opioid utilization and shortens time to full feeding. J Pediatr Surg. 2020 Jan;55(1):101-105. doi: 10.1016/j.jpedsurg.2019.09.065. Epub 2019 Nov 15. PMID 31784102
- [Background] Loganathan AK, Joselyn AS, Babu M, Jehangir S. Implementation and outcomes of enhanced recovery protocols in pediatric surgery: a systematic review and meta-analysis. Pediatr Surg Int. 2022 Jan;38(1):157-168. doi: 10.1007/s00383-021-05008-8. Epub 2021 Sep 15. PMID 34524519